CLINICAL TRIAL: NCT04668612
Title: Lowering Postprandial Hyperglycemia With Dual-wave Insulin Boluses in Children With Type 1 Diabetes
Brief Title: Dual-wave Boluses in Children With Type 1 Diabetes Insulin Boluses in Children With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tartu University Hospital (Other)
Collaborators: Estonian Research Council (Unknown)
Responsible Party: Principal Investigator, Aleksandr Peet, pediatric endocrinologist, MD, PhD, Tartu University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.1
Record Dates: First submitted 2020-11-30; First posted 2020-12-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized open-label single-center crossover clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard-bolus (Active Comparator): Standard boluses for all meal
  Interventions: Device: Standard bolus
- Dual-bolus (Experimental): Dual-bolus (50/50% with second part over 2 hours) for all meals after 6:00 p.m
  Interventions: Device: Dual-bolus

INTERVENTIONS:
Device: Dual-bolus — Dual-bolus (50/50% with second part over 2 hours) for all meals after 6:00 p.m.
  Arms: Dual-bolus
Device: Standard bolus — Standard boluses for all meals
  Arms: Standard-bolus

SUMMARY:
To analyze with the aid of CGM the blood sugar profiles of children receiving dual-wave versus standard bolus for dinner.

DETAILED DESCRIPTION:
Primary objective To analyze with the aid of CGM the blood sugar profiles of children receiving dual-wave versus standard bolus for dinner.

Primary endpoint To compare time in range (TIR) during 2 weeks receiving dual-wave bolus versus standard bolus for dinner.

Trial design This is a 28-day long prospective randomized open-label single-center crossover clinical study with a 14-day long run-in phase.

Trial population A total of 30 subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7-18 years treated at the Children's Clinic of Tartu University Hospital for type1 diabetes.
2. Insulin pump and CGM initiated at least 3 months prior to the recruitment.
3. Estimated HbA1c based on the 14-days CGM report above 8.5%.
4. Daily insulin dose of more than 0.5 international units per kilogram.

Exclusion Criteria:

1. Subjects with known diabetes complications.
2. Elevated tissue transglutaminase IgA antibodies in the last two years.
3. Children who developed an acute viral infections during the week preceding the recruitment.

Exclusion criteria after the Run-in period

1. Basal insulin proportion > 55% of daily insulin dose.
2. Children with any symptoms of an infectious disease or acutely sick during the last two weeks.
3. Estimated HbA1c > 8.5% based on the 14-days CGM report.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) during 2 weeks receiving dual-wave bolus versus standard bolus for dinner. | 14 days
  To compare time in range duration during 2 weeks receiving dual-wave bolus versus standard bolus for dinner. Proportion of time in range (3.9-10 mmol/L) will be measured.

SECONDARY OUTCOMES:
Time below range (TBR) during 2 weeks receiving dual-wave bolus versus standard bolus for dinner. | 14 days
  Time below range (TBR) during 2 weeks receiving dual-wave bolus versus standard bolus for dinner. Proportion of time below range (<3,9 mmol/L)
Time above range (TAR) during 2 weeks receiving dual-wave bolus versus standard bolus | 14 days
  Time above range (TAR) during 2 weeks receiving dual-wave bolus versus standard bolus for dinner. Proportion of time below range (>10.0 mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No